CLINICAL TRIAL: NCT05011864
Title: Integrated Tele-Behavioral Activation and Fall Prevention for Low-income Homebound Older Adults With Depression
Brief Title: Integrated Tele-Behavioral Activation and Fall Prevention for Low-income Homebound Seniors With Depression
Acronym: TBF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Namkee Choi, Professor and Louis and Ann Wolens Centennial Chair in Gerontology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2R01MD009675-07 (NIH)
Record Dates: First submitted 2021-08-06; First posted 2021-08-18 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Depression, Unipolar; Fall
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Intervention Model Description: In a pragmatic RCT design with randomization prior to consent rather than the traditional consent-to-randomization design, we will follow six steps in recruitment, enrollment, and intervention delivery: 1) identification of potential participants by case managers / social workers during in-home or telephone assessments and referral to the research team; 2) randomization into TBF (combined Tele-behavioral activation and fall prevention), Tele-BA, FP, and Attention Control (AC: telephone support calls) arms by the research team; 3) calling each person for consent for telephone eligibility screening; 4) conducting in-depth, in-home screening and baseline assessment for eligible, consenting seniors; 5) delivering TBF, Tele-BA alone, FP alone, or AC; and 6) conducting follow-up assessments.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tele-Behavioral Activation and Fall Prevention (Experimental): Each subject will participate in five 1-hour, weekly Tele-BA sessions followed by four 1-1.5 hour, weekly in-home FP sessions with the same provider
  Interventions: Behavioral: Behavioral Activation; Behavioral: Fall Prevention
- Tele-Behavioral Activation (Experimental): Each subject in this arm will participate in five 1-hour, weekly Tele-BA sessions followed by four weekly check-in (booster) calls of up to 30 minutes each.
  Interventions: Behavioral: Behavioral Activation
- Fall Prevention (Experimental): Each subject will participate in four 1-1.5 hour, weekly in-home (or tele, if COVID continues) FP sessions followed by four weekly check-in (booster) calls of up to 30 minutes each.
  Interventions: Behavioral: Fall Prevention
- Attention Control (Telephone Support Call) (Active Comparator): AC participants in this study will receive five weekly telephone calls of up to 45 minutes each and four weekly check-in calls of up to 30 minutes each from a research assistant (RA) who will employ genuine regard and attentive listening and provide nonspecific support.
  Interventions: Other: Telephone support

INTERVENTIONS:
Behavioral: Behavioral Activation — In BA, depressive symptoms are viewed as depressive behaviors. Compared to those without depression, people with depression engage in fewer overt behaviors that provide positive reinforcement and pleasure/enjoyment and in more behaviors that function to escape or avoid aversive stimuli (e.g., staying in bed all day).55-59 Thus, BA is aimed at increasing and reinforcing meaningful, healthy, and enjoyable behaviors while decreasing depressive behaviors and is well-suited to help depressed, disabled older adults increase mood-enhancing activities, self-care management skills, and social connectedness.
  Other Names: Tele-BA
  Arms: Tele-Behavioral Activation; Tele-Behavioral Activation and Fall Prevention
Behavioral: Fall Prevention — Following FP psychoeducation based on the Centers for Disease Control and Prevention (CDC)'s STEADI tool kits, lay coaches will assist clients in implementing evidence-based FP strategies that have been adapted for low-income homebound seniors. These include referrals to healthcare providers as needed, home safety checks, practice of safe ambulation/transfer and mobility aid use, medication review, and in-home exercise routines with an innovative, gamified tablet-based exercise app for balance and strength building.
  Other Names: FP
  Arms: Fall Prevention; Tele-Behavioral Activation and Fall Prevention
Other: Telephone support — Subjects in this arm will receive 9 weekly support calls last 30 minutes each. These calls are intended to provide an opportunity for social support and check safety.
  Other Names: AC
  Arms: Attention Control (Telephone Support Call)

SUMMARY:
This study will test clinical and cost effectiveness of an integrated tele- and bachelor's-level counselor/coach delivered behavioral activation (BA) and fall prevention (FP) for low-income homebound older adults. The long-term objective of the proposed study is to improve access to depression treatment and fall prevention for growing numbers of low-income homebound seniors. We plan to recruit 320 low-income, racially diverse homebound seniors who are served by a home-delivered meal (HDM) program and other aging-service agencies in Central Texas. In a 4-arm, pragmatic clinical trial with randomization prior to consent, the participants in the integrated Tele-BA and FP (TBF hereafter) arm will receive 5 Tele-BA sessions and 4 in-home FP sessions. Those in the Tele-BA or FP alone arms will receive the respective intervention and 4 bimonthly telephone check-in (booster) calls, and those in the Attention Control (AC) arm will receive 5 weekly telephone check-in calls followed by 4 bimonthly follow-up calls. Follow-up assessments will be at 12, 24, and 36 weeks after baseline.

DETAILED DESCRIPTION:
Depression and falls are significantly higher in low-income, racially diverse homebound seniors than in the general older-adult population; however, the existing systems of care are not equipped to address disparities in mental health and fall prevention services for these vulnerable older adults. The long-term objective of the proposed study is to improve access to depression treatment and fall prevention for growing numbers of low-income homebound seniors. Specific aims are to compare clinical and cost effectiveness of integrated tele-delivered behavioral activation (Tele-BA) and fall prevention (FP) by bachelor's-level lay counselors/coaches to Tele-BA or FP alone and attention control (AC). The current and projected shortages of licensed clinicians and the costs of deploying highly trained professionals pose barriers to providing services to older adults in general and low-income homebound seniors in particular. A more scalable option is to utilize lay counselors/coaches, and our recent clinical trial (1R01MD009675) and a FP pilot study show that lay counselors/coaches are as effective as licensed clinicians. The study participants will be 320 low-income, racially diverse homebound seniors who are served by a home-delivered meal (HDM) program and other aging-service agencies in Central Texas. The lay counselors/coaches will be co-located in the HDM program for seamless referral and care coordination. In a 4-arm, pragmatic clinical trial with randomization prior to consent (a preferred public health approach), the participants in the integrated Tele-BA and FP (TBF hereafter) arm will receive 5 Tele-BA sessions and 4 in-home FP sessions. Those in the Tele-BA or FP alone arms will receive the respective intervention and 4 bimonthly telephone check-in (booster) calls, and those in the AC arm will receive 5 weekly telephone check-in calls followed by 4 bimonthly follow-up calls. Study hypotheses are: At 12, 24, and 36 weeks after baseline, (1) TBF will be more effective than Tele-BA or FP alone, and Tele-BA or FP alone will be more effective than AC in reducing depression (the 24-item Hamilton Rating Scale for Depression), falls, and fall injuries; (2) TBF than Tele-BA alone or FP alone will be more effective in reducing disability (WHODAS 2.0) and healthcare and social service use; and (3) TBF will be more cost effective than Tele-BA alone or FP alone. Cost-effectiveness analysis (CEA) will be based on depression free days, prevented falls, and health-related quality adjusted life-year measured by EuroQol-5 (EQ-5D). We will also conduct budget impact analysis (BIA) of TBF relative to Tele-BA or FP. Both CEA and BIA will employ a hybrid public program perspective of the Administration for Community Living and the Centers for Medicare and Medicaid. Public health significance of this study is that it will provide empirical data needed for real-world adoption of an intervention delivery model that targets to intervene for the two most frequent sources of disability acceleration and healthcare use among a rapidly growing, underserved population. (We use the terms older adults and seniors interchangeably because the latter term is frequently used in aging services.)

ELIGIBILITY:
Inclusion Criteria:

* Age 50+
* English or Spanish proficiency
* 24-item Hamilton Rating Scale for Depression score > 15
* 12-item Fall Risk Questionnaire score >4

Exclusion Criteria:

* Recently (< 4 weeks) initiated or modified antidepressant pharmacotherapy
* High suicide risk
* Probable dementia
* Bipolar disorder
* Substance use/misuse
* Current participation in any psychotherapy or FP program
* Bedbound status

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline depressive symptom at 12, 24, and 36 weeks | at 12, 24, and 36 weeks after baseline
  24-item Hamilton Rating Scale for Depression score (score range: 15-40; decreased score since baseline is a positive outcome)
Changes from baseline fall count and injury at 12, 24, and 36 weeks | monthly (form 12 weeks to 36 weeks)
  Changes in six monthly falls calendar data (reduced number of falls since baseline is a positive outcome)
Changes from baseline EuroQol-5D score at 12, 24, and 36 weeks | at 12, 24, and 36 weeks after baseline
  Cost-effectiveness measure (score range: 0-20; decreased score since baseline is a positive outcome)
Changes from baseline physical and mental health service use | at 12, 24, and 36 weeks after baseline
  Changes in Cornell Services index data (decreased ED visits and hospitalization since baseline is a positive outcome)
Changes from baseline disability score at 12, 24, and 36 weeks | at 12, 24, and 36 weeks after baseline
  Changes in 12-item World Health Organization Disability Assessment Schedule score (score range: 0-46; decreased score since baseline is a positive outcome)
Changes from baseline social engagement and activities score at 12, 24, and 36 weeks | at 12, 24, and 36 weeks after baseline
  Changes in 10-item Social Engagement and Activities Questionnaire score (score range: 0-50; increased score since baseline is a positive outcome)
Changes from baseline satisfaction with social roles & activities at 12, 24, and 36 weeks | at 12, 24, and 36 weeks after baseline
  C (score range: 0-32; increased score since baseline is a positive outcome)

SECONDARY OUTCOMES:
Changes from baseline fear of falling at 12, 24, and 36 weeks | at 12, 24, and 36 weeks after baseline
  Changes in 7-item Falls Efficacy Scale International score (score range: 7-28; decreased score since baseline is a positive outcome)
Changes from baseline exercise frequency at 12, 24, and 36 weeks | at 12, 24, and 36 weeks after baseline
  Changes in RAPA (Rapid Assessment of Physical Activities) (score range: 1-9; increased score since baseline is a positive outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Namkee G Choi, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No